CLINICAL TRIAL: NCT03209635
Title: Weissella Cibaria JW15 Consumption and NK Cell Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, Yonsei University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: AI_probiotic_NK
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Immune Function
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 4 capsules (300 mg/capsule) containing 52% crystalline cellulose and 46% lactose in identical-looking with test product
  Interventions: Dietary Supplement: Placebo
- Probiotic (Experimental): 4 capsules (300 mg/capsule) containing each capsule 1.0 x 10^10 colony-forming units (cfu) of Weissella cibaria JW15, twice a day
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Placebo — 4 capsules (300 mg/capsule) containing 52% crystalline cellulose and 46% lactose in identical-looking with test product
  Arms: Placebo
Dietary Supplement: Probiotic — 4 capsules (300 mg/capsule) containing each capsule 1.0 x 10^10 colony-forming units (cfu) of Weissella cibaria JW15, twice a day
  Arms: Probiotic

SUMMARY:
A The aim of this study was to investigate the impact of consuming Weissella cibaria (W. cibaria) JW15 supplementation isolated from Kimchi, Korea traditional fermented food, on natural killer (NK) cell activity and circulating levels of cytokines and immunoglobulin (Ig).

DETAILED DESCRIPTION:
A randomized, double-blinded, placebo-controlled study was conducted on 100 nondiabetic subjects. Over an eight-week testing period, the probiotic group consumed 4 capsules (300 mg/capsule) containing 1 x 10^10 colony-forming units (cfu) of W. cibaria JW15 each day, whereas the placebo group consumed the same product without a probiotic.

ELIGIBILITY:
Inclusion Criteria:

* Nondiabetic (fasting serum glucose concentration < 126 mg/dL)
* Subjects with 4,000-8,000 leukocyte counts

Exclusion Criteria:

* Constant consumption of any probiotic products
* Taking medicine related to inflammation within one month before screening
* Allergy to probiotics
* Lactose intolerance
* Diabetes
* History/presence of significant metabolic disease
* Acute or chronic disease requiring treatment
* Taking any medications

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Natural killer cell activity at baseline | Baseline
  Natural killer cell activity (%)
Natural killer cell activity at 8-week follow up | 8-week follow up
  Natural killer cell activity (%)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D., Principal Investigator — Dept. of Food and Nutrition, Colleage of Human Ecology, Yonsei University

IPD SHARING:
Plan to Share IPD: No